CLINICAL TRIAL: NCT00376259
Title: An Open-label, Multicenter, Randomized Study of Combination Therapy With Oral LDT600 (Telbivudine) Plus Adefovir Dipivoxil Versus Adefovir Dipivoxil Alone in HBeAg-positive Patients With Chronic Hepatitis B Who Are Lamivudine Resistant
Brief Title: Study of Combination Therapy With LdT Plus Adefovir Versus Adefovir Alone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not completed as planned and was terminated early with agreement from the European Medicines Agency (EMEA)
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2304
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis B
Keywords: lamivudine resistance; Hepatitis B virus
MeSH Terms: conditions — Hepatitis B | interventions — Telbivudine; adefovir dipivoxil

ARMS (2):
- Combination therapy (Experimental): Combination therapy: 600 mg of telbivudine (LdT) by mouth plus 10 mg of adefovir (ADV) by mouth once daily for 96 weeks.
  Interventions: Drug: telbivudine; Drug: adefovir dipivoxil
- Adefovir monotherapy (Active Comparator): Adefovir monotherapy: 10 mg of adefovir by mouth once daily for 96 weeks.
  Interventions: Drug: adefovir dipivoxil

INTERVENTIONS:
Drug: telbivudine — 600mg/day oral tablet for 96 weeks
  Arms: Combination therapy
Drug: adefovir dipivoxil — 10 mg of adefovir by mouth once daily

SUMMARY:
This study is being conducted to compare the safety and effectiveness of the investigational medication LdT (telbivudine) used in combination with adefovir dipivoxil (a drug currently approved by the Food and Drug Administration [FDA] for the treatment of hepatitis B virus [HBV]) versus adefovir dipivoxil used alone. The results for patients taking the combination therapy will be compared to the results for patients taking adefovir alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented compensated chronic hepatitis B defined by a clinical history compatible with chronic hepatitis B.
* Previous or current lamivudine treatment
* HBV DNA > 6 log10 copies/mL
* Evidence of viral breakthrough

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Patient is pregnant or breastfeeding.
* Patient is co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV.
* Patient has received any anti-HBV treatment for HBV infection other than lamivudine in the 12 months before Screening for this study.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Novartis, San Diego, California
  - San Mateo, California
- Pok Fu Lam, Hong Kong
- Seoul, South Korea
- Novarits, Kaohsuing, Taiwan
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment was 150 patients. At the time of study termination, 43 patients had been enrolled and randomized to study treatment and 42 patients received study drug (21 patients in the combination group and 21 in the monotherapy group).
Pre-assignment Details: One patient was randomized but never received study drug treatment because he was discontinued on the randomization day due to sponsor request.
Period: Overall Study
Arm/Group | Combination Therapy | Adefovir Monotherapy
Started | 22 | 21
Received Study Drug | 21 | 21
Completed | 0 | 0
Not Completed | 22 | 21
Not completed — Sponsor request - study termination | 21 | 21
Not completed — Patient request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Adefovir Monotherapy | Total
Number analyzed (Participants) | 22 | 21 | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.82) | 39.0 (10.93) | 37.9 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 19 | 16 | 35

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Experienced Virologic Breakthrough
Description: Virologic breakthrough is defined as a minimum of 1 log reduction from baseline followed by a 1 log increase from nadir on at least 2 consecutive visits including the last treatment visit.
Time Frame: 96 Weeks
Population: This study was terminated early and no patients received 96 weeks of treatment. Therefore, the primary objective of evaluating virologic breakthrough by Week 96 could not be assessed. Consequently, all protocol-specified inferential analyses on the primary endpoint and all other key secondary efficacy endpoints could not be performed.
Measure: Number; unit: Proportion of participants
Arm/Group | Combination Therapy | Adefovir Monotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Mean Hepatitis B Virus (HBV) DNA Concentration
Description: Efficacy was assessed by the change from baseline in mean HBV DNA concentration after 12, 24, 48 and 60 weeks of treatment.
Time Frame: Baseline to 12 weeks, 24 weeks, 48 weeks and 60 weeks
Population: Analysis population consists of the intent-to-treat population. Analysis of data for each time point includes participants who had both baseline and post baseline observation.
Measure: Mean (Standard Deviation); unit: Log10 Copies/mL
Arm/Group | Combination Therapy | Adefovir Monotherapy
Number analyzed (Participants) | 21 | 21
Log10 Copies/mL
  At Baseline (N = 21, 20) | 10.240 (1.5750) | 10.127 (0.9697)
  At Week 12 | 4.405 (0.9944) | 5.515 (1.3188)
  Change from Baseline to Week 12 | -5.835 (1.6435) | -4.612 (1.7725)
  At Baseline (N = 20, 20) | 10.279 (1.6058) | 10.127 (0.9697)
  At Week 24 | 3.678 (1.0483) | 5.161 (1.7364)
  Change from Baseline to Week 24 | -6.601 (1.7873) | -4.966 (2.2851)
  At Baseline (N = 13, 9) | 10.652 (1.5203) | 10.207 (0.7520)
  At Week 48 | 3.274 (1.0254) | 5.272 (1.9581)
  Change from Baseline to Week 48 | -7.378 (1.9303) | -4.934 (2.1153)
  At Baseline (N = 2, 3) | 9.605 (0.7990) | 10.097 (0.1484)
  At Week 60 | 3.360 (0.3111) | 4.330 (0.6110)
  Change from Baseline to Week 60 | -6.245 (0.4879) | -5.767 (0.4650)

3. Secondary Outcome: Percentage of Participants Achieving Specified Clinical and Laboratory Safety Criteria
Description: Undetectable HBV DNA = HBV DNA <300 copies/ml. Serum aminotransferase (ALT) normalization is defined as ALT within normal limits on 2 successive visits for a pt. with an elevated ALT level (>=1.0 x ULN) at baseline (BL). Hepatitis B e antigen (HBeAg) loss is defined as the loss of detectable serum HBeAg in a pt. who was HBeAg +ve at BL. HBeAg seroconversion is defined as HBeAg loss with detectable HBeAb. Hepatitis B surface antigen (HBsAg) loss is defined as the loss of detectable serum HBsAg in a pt. who was HBsAg +ve at BL. HBsAg seroconversion is defined as HBsAg loss with detectable HBsAb.
Time Frame: 12 week, 24 week, 48 week and 60 weeks
Population: Analysis population consists of the intent-to-treat population. Analysis of data for each time point includes participants who had both baseline and post baseline observation for that timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Combination Therapy | Adefovir Monotherapy
Number analyzed (Participants) | 21 | 21
Percentage of participants
  Undetectable HBV DNA at week 12 | 4.8 | 5.0
  Undetectable HBV DNA at week 24 | 15.0 | 10.0
  Undetectable HBV DNA at week 48 | 38.5 | 0.0
  Undetectable HBV DNA at week 60 | 0.0 | 0.0
  Serum ALT normalization at week 12 | 40.0 | 25.0
  Serum ALT normalization at week 24 | 55.0 | 35.0
  Serum ALT normalization at week 48 | 69.2 | 33.3
  Serum ALT normalization at week 60 | 50.0 | 0.0
  HBeAg loss at week 12 | 0.0 | 0.0
  HBeAg loss at week 24 | 5.0 | 5.0
  HBeAg loss at week 48 | 23.1 | 0.0
  HBeAg loss at week 60 | 0.0 | 0.0
  HBeAg seroconversion at week 12 | 0.0 | 0.0
  HBeAg seroconversion at week 24 | 0.0 | 0.0
  HBeAg seroconversion at week 48 | 15.4 | 0.0
  HBeAg seroconversion at week 60 | 0.0 | 0.0
  HBsAg loss at week 12 | 0.0 | 0.0
  HBsAg loss at week 24 | 0.0 | 0.0
  HBsAg loss at week 48 | 0.0 | 0.0
  HBsAg loss at week 60 | 0.0 | 0.0
  HBsAg seroconversion at week 12 | 0.0 | 0.0
  HBsAg seroconversion at week 24 | 0.0 | 0.0
  HBsAg seroconversion at week 48 | 0.0 | 0.0
  HBsAg seroconversion at week 60 | 0.0 | 0.0

4. Secondary Outcome: Proportion of Participants With Treatment-emergent HBV Resistance Mutations Associated With Virologic Breakthrough
Description: The study was not completed as planned and was terminated early with agreement from the European Medicines Agency (EMEA). Patients did not receive 96 weeks of treatment. Therefore, the primary objective of evaluating virologic breakthrough by Week 96 could not be assessed. Consequently, all protocol-specified inferential analyses on the primary endpoint and all other key secondary efficacy endpoints could not be performed.
Time Frame: Week 96
Measure: Number; unit: Proportion of Participants
Arm/Group | Combination Therapy | Adefovir Monotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Safety population.
Arm/Group | Combination Therapy | Adefovir Monotherapy
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21
Other Adverse Events (participants affected / at risk) | 14/21 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=21) | Adefovir Monotherapy (N=21)
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy (N=21) | Adefovir Monotherapy (N=21)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 3
Hepatic steatosis (Hepatobiliary disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0
Rhinitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 8
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was not completed as planned and was terminated early with agreement from the European Medicines Agency (EMEA).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.